CLINICAL TRIAL: NCT03850171
Title: Importance of Exercise Training Therapy Timing With Regard to Cardiotoxicity and Patient Preference in Early Breast Cancer and Lymphoma Patients Undergoing Adjuvant Chemotherapy
Brief Title: Cancer Adverse Effects PReventIon With Care & Exercise: the CAPRICE Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the lack of financial and human resources the investigators were unable to continue the study. The targeted sample size was not achieved due to recruitment difficulties (mainly related to the Covid-19 pandemic).
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Spital STS AG (Industry); Bürgerspital Solothurn (Other); Lindenhofspital (Unknown); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAPRICE
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Breast Neoplasm Female; Lymphoma; Cardiotoxicity; Anthracyclines; Physical Activity
Keywords: Breast Cancer; Exercise Training Therapy; Global longitudinal strain; Barriers; Left ventricular dysfunction; Heart failure; Breast disease; Exercise rehabilitation; Lymphoma
MeSH Terms: conditions — Lymphoma; Cardiotoxicity; Motor Activity; Breast Neoplasms; Ventricular Dysfunction, Left; Heart Failure; Breast Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised, controlled; parallel arm design.
Who Masked: Outcomes Assessor
Masking Description: Assessors of outcome data and analysis will be blinded to the intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ExEarly (Experimental): Patients completing the exercise training concurrent to anthracycline chemotherapy treatment during months 1 to 3
  Interventions: Other: Exercise Training
- ExStandard (No Intervention): Patients will be encouraged to continue with their regular physical activity routine and will be medically managed as per standard of care by their Cardiologist and Oncologists.

INTERVENTIONS:
Other: Exercise Training — Participants from the experimental study arm are assigned to a 12-week exercise training programme integrated in a multidisciplinary oncology rehabilitation programme at the Inselspital Bern, Spital AG Thun, or Bürgerspital Solothurn. The exercise programme will comprise 2 weekly exercise sessions lasting 90 min, supervised by experienced exercise therapists. The sessions start with approximately 40 min cycling on an ergometer at moderate intensity, increasing on a weekly basis if possible. After the cycling training, patients continue the exercise session with 40 min of strength training, stretching, relaxation, coordination and balance training. In addition, patients will be instructed to perform at least one additional endurance-related activity per week in their own time with a duration of 30-60 min at moderate intensity levels (e.g. walking, bicycling).
  Arms: ExEarly

SUMMARY:
Breast cancer is the most common cancer among women worldwide. Similarly, Hodgkin and non- Hodgkin lymphomas make up two of the most prevalent cancers in men and women. Even though remarkable improvements in cancer-free survival have been achieved in the last decades, the development of cardiac toxicity, associated with anthracycline-based chemotherapy (Anth-bC) counteracts the improvements in survival in these patient groups. One of the first clinical manifestation of Anth-bC cardiotoxicity is diastolic dysfunction, with further symptoms being left ventricular dysfunction and heart failure as well as a decline in exercise tolerance. Besides the direct cardiotoxic effects of anticancer treatment, many drugs also have adverse effects on the vascular endothelium.

The concept of 'Exercise is Medicine' has become well established in exercise-oncology research. Exercise therapy is now considered a safe and well-tolerated adjunct therapy inducing beneficial effects on body composition, aerobic fitness and muscular strength, pain and fatigue, quality of life (QoL), depressive symptoms, and all cause survival. However, there is insufficient data on the superiority of performing exercise training therapy before and during chemotherapy with regard to cardiotoxic and cardiovascular side effects. Further, there is no data on patient preference for and barriers toward different timings of exercise training therapy.

Therefore, the aim of the study is to compare left ventricular (LV) function measured by LV global longitudinal strain (GLS) in breast cancer and lymphoma patients undergoing Anth-bC randomised to completing an exercise-based rehabilitation programme during chemotherapy to those randomised to complete the programme after chemotherapy. Further, blood samples will be drawn to analyse biomarkers of myocardial injury (brain natriuretic peptide and high-sensitive cardiac troponin).

Additional measurements include aortic distensibility as part of the echocardiographic examination and exercise capacity through cardiopulmonary exercise testing. QoL and fatigue will be assessed in a questionnaire, compliance with exercise training through monitoring and patient preference at 3 and 6 months will be evaluated through an interview. Cardiovascular risk factors will be assessed through body composition, 24h ambulatory blood pressure monitoring, 24h electrocardiogram and the analysis of established blood markers.

Women and men aged 18 years and older with histologically confirmed breast cancer or lymphoma (ECOG grade 0-2) who are Anth-bC naïve and with reasonable life expectancy will be included in the study.

The exercise programme is part of onco-rehabilitation programmes at the Inselspital Bern, the Spital AG Thun and the Bürgerspital Solothurn. Programmes last for 12 weeks and offer two supervised sessions per week (@ 60-90 min). They usually contain an endurance component (e.g. 40 min of cycling) and a strength, agility or relaxation component. Patients are encouraged to complete a third exercise session per week at home or elsewhere. Home-based training and general physical activity will be assessed by a questionnaire and an activity monitor.

A total of 120 patients will be recruited. Measurements will be performed at baseline, after 3 months (week 13) and after 6 months (week 26).

DETAILED DESCRIPTION:
Study Design: A single-center, two-arm, parallel group with standard of care controlled trial with a balanced 1:1 randomization will be conducted at University Hospital Inselspital, Berne, Switzerland. A total of 120 women (60 participants per study arm) who are scheduled for first- line Anthracycline based chemotherapy (Anth-bc) presenting either at the Inselspital or Lindenhofspital Berne, the Spital AG Thun or the Bürgerspital Solothurn will be enrolled. After baseline assessments, eligible participants will be randomized to one of two arms including the exercise rehabilitation programme during chemotherapy or the control group (exercise training intervention after conclusion of chemotherapy).

Patient Population: Women and men aged 18 years and older with histologically confirmed breast cancer or lymphoma who are Anth-bC naïve and are scheduled for first-line Anth-bC, Eastern Cooperative Oncology Group (ECOG) grade 0-2, curative or palliative approach with reasonable life expectancy and a willingness to attend exercise sessions twice per week for 12 weeks (24 sessions in total).

Procedures: The following measurements will be collected at the beginning (T0), following the 12 week intervention (T1) and after another 12 weeks (T2). Participants will also be expected to attend two weekly supervised exercise sessions integrated in a multidisciplinary oncology rehabilitation programme at the Inselspital Bern, Spital AG Thun, and Bürgerspital Solothurn, and will be expected to complete one additional exercise training session at home or in the community each week.

T0: All participants will undergo baseline assessments at the University Hospital Inselspital, Berne. This includes cardiac assessment by a skilled clinical cardiac sonographer to obtain left ventricular (LV) global longitudinal strain (GLS) and aortic distensibility. Further, cardiopulmonary exercise testing (CPET) will be completed on a cycle ergometer to obtain VO2peak and to calculate corresponding training zones. Standard measures conducted during the intake process including height, weight, body composition (assessed by bio-impedance- measurement) and waist circumference will also be collected. Blood samples will be obtained from each participant and analyzed for biomarkers of myocardial injury as well as lipid profile and HbA1C. Following each visit, twenty-four-hour ambulatory blood pressure monitoring and 24h Holter ECG will be performed. The questionnaires for physical activity patterns (GPAQ) and fatigue (FACIT-F), a health history questionnaire and the activity tracking devices will also be administered by the research coordinator upon their initial visit.

T1: All measurements from T0 will be repeated. Additionally, patients from the ExEarly (experimental) group will be interviewed by the study coordinator to assess barriers for missed exercise sessions. Simultaneously, patients from the ExStandard group will be asked to anticipate barriers which may impede their participation in regular exercise training during the next 12 weeks. It will further be assessed whether it would have been feasible for them to complete the exercise programme concurrently to chemotherapy.

T2: All measurements from T0 will be repeated. Additionally, patients from the ExStandard (active comparator) group will be interviewed by the study coordinator to assess barriers for missed exercise sessions. Simultaneously, patients from the ExEarly group will be asked to indicate their preferred time point for the completion of the exercise programme.

Throughout the programme: Information regarding adherence to the exercise programme will also be collected by the research coordinator each month via the exercise training diaries and activity tracking devices from each participant. The study coordinator will also assess reasons for missed exercise sessions. Lastly, chemotherapy adherence will be assessed by dose adjustments in percent of the intended dose and reason for adjustment.

Intervention (ExEarly): The 12-week exercise training programme will be integrated in a multidisciplinary oncology rehabilitation programme at the Inselspital Bern, Spital AG Thun, and Bürgerspital Solothurn. The exercise programme will comprise 2 weekly exercise sessions lasting 90 min, supervised by experienced exercise therapists. The sessions start with approximately 40 min cycling on an ergometer at moderate intensity, increasing on a weekly basis if possible. After the cycling training, patients continue the exercise session with 40 min of strength training, stretching, relaxation, coordination and balance training. In addition, patients will be instructed to perform at least one additional endurance-related activity per week in their own time with a duration of 30-60 min at moderate intensity levels (e.g. walking, bicycling). In the ExEarly group, patients start in the week preceding the first dose of Anth-bC. They perform exercise training therapy for 12 weeks during which they will normally have 4 cycles of Anth-bC.

Control Group (ExStandard): Participants who are randomized to the control group will undergo baseline and follow up assessments at 13 and 26 weeks. They will be encouraged to continue with their regular physical activity routine and will be medically managed as per standard of care by their Cardiologist and Oncologists. All participants will also complete the GPAQ Questionnaire to determine if there are potential increases in physical activity in the exercise and control group, which may account for changes in all outcome measures. 1-4 weeks after completion of their last dose of Anth-bc the participants will commence exercise training. All participants in both groups will also be asked to wear an activity-tracking device, namely a step counter (Fitbit Zip) during the intervention and control period (25 weeks) to objectively quantify their daily physical activity.

Randomization: Randomization will occur at the central site, the University Hospital, Inselspital Berne, using minimisation based on strata recruiting center, age, therapy (adjuvant/ neoadjuvant), Global Longitudinal Strain (GLS), HER2 status and metastases, with an allocation ratio of 1:1.

Blinding: The participants will not be blinded to their intervention arm. Assessors of outcome data and analysis will be blinded to the study arm.

Analytical Plan: The primary outcome, change in global longitudinal strain (GLS) from before Anth-bC to immediately after Anth-bC (T1 vs T0), will be compared between the two groups (ExEarly and ExStandard) by independent one-sided t-test (or Wilcoxon two-sample test as appropriate) with alpha set at 0.05. Values from baseline (before Anth-bC, T0), completion of Anth-bC (week 13, T1), and follow-up (T2) will be compared between groups using ANCOVA with repeated measures (or mixed models in case of missing data) including baseline values as covariate and post-hoc testing for different time points. Intention-to-treat (ITT) analysis will be performed with group allocation according to randomization to assess the effectiveness of ExEarly in the clinical setting. Per-protocol analysis will be performed with patients allocated with regard to time period they completed more supervised sessions in, with a minimum requirement of 15 of the 24 (60%) scheduled training sessions within one or the other time period to assess the potential effects of an optimal training. Linear models will be performed to find independent baseline parameters to predict negative outcome of cardiac function (LV GLS, NT-proBNP, hsTnT). Secondary endpoints will be analysed accordingly. Statistical analyses will be performed using the software R (Version 3.3.1, R Core Team, 2016).

Significance: Outcomes from this project will improve long term care of patients with early breast cancer and lymphoma as well as other cancers, such that patients can be offered the possibility of active involvement towards mitigating undesirable side effects of a very effective cancer treatment. The assessment of barriers to training therapy may help to adapt the offered physical training programmes to reduce these barriers.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 years and older
* Histologically confirmed breast cancer or lymphoma
* Anth-bC naïve
* Scheduled for first-line Anth-bC
* Eastern Cooperative Oncology Group (ECOG) grade 0-2
* Curative or palliative approach with reasonable life expectancy
* Willingness to attend exercise sessions twice per week for 12 weeks (24 sessions in total)
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Inability to participate in a 3-month training program
* Contraindication to maximal CPET
* Cancer-specific contraindications including safety blood parameters
* Previous radiotherapy of the mediastinum and/or the the left breast
* Structural heart disease with reduced left ventricular ejection fraction (EF<50%)
* Valvular heart disease with more than mild regurgitation or stenosis
* Heart rhythms other than sinus rhythm
* Pacemaker with permanent ventricular stimulation
* Antihypertensive medication (e.g. ACE inhibitors/ATII blockers, Ca channel blocker, beta blockers)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in left ventricular (LV) global longitudinal strain (GLS) | week 13
  GLS assessed by speckle tracking echocardiography is an established marker for LV systolic function with a good reproducibility, which has also been found in the investigators' laboratory. In breast cancer and lymphoma patients LV global longitudinal strain is an established measure to assess cardiotoxicity of Anth-bC.

SECONDARY OUTCOMES:
Change in Blood biomarkers | week 0, 13, and 26
  Blood samples will be collected to determine concentration of Brain Natriuretic Peptide (NT- proBNP) and high- sensitive cardiac Troponin (hsTnT). Cardiac troponin release after high-dose chemotherapy is a marker for chemotherapy-induced cardiotoxicity in cancer patients and identifies patients at different risks of cardiac events in the years thereafter. The increment of hs-TnT has been found to be predictive for cardiotoxicity in breast cancer patients at 3 months after initiation of Anth-bC. Both, NT-proBNP and hs-TnT have been recommended as early biomarkers of cardiotoxicity by the European Society of Cardiology in the guidelines on cancer treatments and cardiovascular toxicity.
Identification of barriers towards exercise training | week 13 and 26
  Barriers toward exercise training therapy will be identified by a self-designed questionnaire.
Compliance with exercise training | week 0, 13 and 26
  Number of attended center-based sessions will be monitored by the attending physiotherapists. Additional home-based training and general physical activity will be assessed by the GPAQ- questionnaire. It collects information on physical activity participation in three domains (work, transport and recreational activities) as well as sedentary behaviour, comprising 16 questions (P1-P16). Within the work and discretionary domains, questions assess the frequency and duration of activity defined by the energy requirement or intensity (vigorous- or moderate-intensity). In the transport domain, the frequency and duration of all walking and cycling for transport is captured. The main outcome variables from GPAQ analysis include a categorical variable of total physical activity (high, moderate and low) and a continuous variable of total physical activity within each domain (reported as Median METmin/week), which will be used to quantify the volume of weekly physical activity.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | week 0, 13, and 26
  The FACIT-F (version 4.0) is a 41-item compilation of general questions divided into four domains of cancer-specific quality of life (physical well-being ranging from 0-28, social/family well-being ranging from 0-28, emotional well-being ranging from 0-24 and functional well-being ranging from 0-28) and a module for fatigue (13 items, ranging from 0- 52).FACIT-F total score ranges from 0- 160. It is considered appropriate to use in patients with any form of cancer. This questionnaire has been validated and used extensively, including reference data for clinically meaningful changes. Change in fatigue will be tested as primary quality of life endpoint.
Vascular function | week 0, 13, and 26
  Vascular function will be assessed by distensibility of the ascending aorta measured on the echocardiography. This is an established measure of arterial stiffness and has recently been shown to decrease from before to after Anth-bC in women with breast cancer. Increased arterial stiffness has been proposed to increase LV afterload, which may lead to LV hypertrophy and in its worst case LV failure.
Cardiorespiratory fitness | week 0, 13, and 26
  Cardiopulmonary exercise testing (CPET) will be performed on a cycle ergometer according to the recommendations of the American Heart Association. VO2peak has been found to be reduced after chemotherapy. It is an established marker for physical function and survival.
Cardiovascular risk profile | week 0, 13, and 26
  It has been suggested that the presence of cardiovascular risk factors increase the risk of developing Anth-bC associated cardiac dysfunction. Twenty-four-hour ambulatory blood pressure monitoring will be performed using validated recorders (Spacelabs model 90217, USA) during usual daily activities. Lipid profile and HbA1C will be determined from blood samples. Body composition will be measured by bio-impedance measurement (InBody 720, Biospace Co., Seoul, Korea) and smoking status will be assessed. Also, a 24-hour Holter electrocardiogram will be performed. Both 24-hour monitors will be worn after each visit on two separate days.
Changes in LV global longitudinal strain | Week 0 and 26
  GLS assessed by speckle tracking echocardiography is an established marker for LV systolic function with a good reproducibility, which has also been found in the investigators' laboratory. In breast cancer and lymphoma patients LV global longitudinal strain is an established measure to assess cardiotoxicity of Anth-bC.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Wilhelm, Prof. Dr., Principal Investigator — University Clinic for Cardiology, University Hospital Berne
Locations (4):
- Switzerland (4):
  - Lindenhofgruppe, Bern
  - University Clinic for Cardiology, Bern
  - Bürgerspital Solothurn, Solothurn
  - Spital STS AG, Thun

IPD SHARING:
Plan to Share IPD: Yes
Upon request, de-identified individual participant data for research purposes will be made available as far as legally permissible.

REFERENCES:
- [Derived] Schneider C, Ryffel C, Stutz L, Rabaglio M, Suter TM, Campbell KL, Eser P, Wilhelm M. Supervised exercise training in patients with cancer during anthracycline-based chemotherapy to mitigate cardiotoxicity: a randomized-controlled-trial. Front Cardiovasc Med. 2023 Dec 4;10:1283153. doi: 10.3389/fcvm.2023.1283153. eCollection 2023. PMID 38111886